CLINICAL TRIAL: NCT06005727
Title: Cryotherapy Post-haemorrhoidectomy (CYPHER) Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/2357
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Hemorrhoids; Postoperative Pain; Postoperative Complications; Cryotherapy Effect
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transanal ice pack applied to hemorrhoidectomy wound for 1 minute (Active Comparator): Transanal ice pack is applied to hemorrhoidectomy wound for 1 minute. After the surgery, standard postoperative analgesia and medications will be prescribed.
  Interventions: Device: Transanal ice pack
- Standard postoperative care after hemorrhoidectomy (No Intervention): Standard postoperative analgesia and medications will be prescribed.

INTERVENTIONS:
Device: Transanal ice pack — A condom is filled with 100ml of water and frozen to serve as a transanal ice pack. It is covered by sterile plastic dressing and applied to the hemorrhoidectomy wound for 1 minute after surgery is completed.
  Arms: Transanal ice pack applied to hemorrhoidectomy wound for 1 minute

SUMMARY:
Haemorrhoids is a common problem with an estimated prevalence of 5 to 36%. Surgery is indicated in patients with grade 3 to 4 piles and in patients whom conservative measures have failed. There have been several surgical techniques described such as the Milligan- Morgan, Ferguson haemorrhoidectomy, stapled and laser haemorrhoidectomy. However, most patients experience different degrees of postoperative pain which may cause anxiety and dissatisfaction.

A relatively non-invasive and cost-effective technique targeting inflammation is cryotherapy which has been shown to decrease pain secondary to trauma, injury or disease. Cryotherapy has few deleterious side effects due to its non-pharmacologic nature and has become widespread in sports medicine to treat soft tissue damage.

Therefore, we aim to evaluate the role of cryotherapy in improving postoperative pain and outcomes among patients who undergo haemorrhoidectomy.

DETAILED DESCRIPTION:
Haemorrhoids is a common problem with an estimated prevalence of 5 to 36%. Surgery is indicated in patients with grade 3 to 4 piles and in patients whom conservative measures have failed. There have been several surgical techniques described such as the Milligan- Morgan, Ferguson haemorrhoidectomy, stapled and laser haemorrhoidectomy. However, most patients experience different degrees of postoperative pain which may cause anxiety and dissatisfaction.

Pain is an unavoidable side effect of any proctology operation. It arises from local inflammation in traumatized tissues which may cause stimulation of surrounding nociceptors. While adequate postoperative analgesia promotes patient recovery and satisfaction, narcotics for postoperative pain are also associated with numerous side effects.

A relatively non-invasive and cost-effective technique targeting inflammation is cryotherapy which has been shown to decrease pain secondary to trauma, injury or disease. Cryotherapy has few deleterious side effects due to its non-pharmacologic nature and has become widespread in sports medicine to treat soft tissue damage. Ice therapy has previously been shown to be safe and effect for postoperative analgesia in various procedures such as laparotomy, hernia repair, tonsillectomy, oral surgery but the evidence for its role in haemorrhoidectomy is lacking.

Therefore, we aim to evaluate the role of cryotherapy in improving postoperative pain and outcomes among patients who undergo haemorrhoidectomy. We hypothesize that intraoperative trans-anal ice pack insertion for patients after haemorrhoidectomy (conventional & stapled) will have lower postoperative pain scores with possibly decreased postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age group of patients: 21 to 75 years old
2. Grade 3 (prolapsed but reducible manually) and Grade 4 (prolapsed but irreducible) piles that are symptomatic
3. Patients recruited are to undergo either staple or conventional (Milligan-Morgan or Ferguson) haemorrhoidectomy

Exclusion Criteria:

1. Grade 1 and 2 haemorrhoids
2. Thrombosed, irreducible piles that require emergency haemorrhoidectomy
3. Patients who had undergone any previous anorectal surgery within 5 years from the date of recruitment
4. Patients with concurrent anorectal pathology (anal fissures, abscess, fistula, tumour, inflammatory bowel disease)
5. Pregnant women
6. Patients with severe medical comorbidities or assessed as ASA 3 and above
7. Patients on long term antiplatelets (aspirin, plavix) and anticoagulation (clexane, warfarin, rivaroxaban, apixaban)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score on postoperative day 1 after hemorrhoidectomy | Postoperative day 1
  Pain score on postoperative day from scale of 1 to 10 after hemorrhoidectomy.

SECONDARY OUTCOMES:
Postoperative complications after hemorrhoidectomy | Within 30 days after surgery
  Postoperative bleeding, urinary retention, perianal sepsis, anal stenosis, incontinence
Proportion of patients who had admission after day surgery or readmission for postoperative complications | Within 30 days after surgery
  Proportion of patients who had readmission or required admission after surgery.
Proportion of patients who require repeat surgical interventions for postoperative complications: bleeding, perianal sepsis and anal stenosis | Within 30 days after surgery
  Proportion of patients who required repeat surgical interventions after surgery.
Changes in the mean pain score 1 month after surgery assessed by telephone interviews on POD1, 2, 3, 4, 7, 14, 21 and 28. | Postoperative day 1, 2, 3, 4, 7, 14, 21 and 28.
  Pain scores are recorded on the postoperative day 1, 2, 3, 4, 7, 14, 21 and 28 and postoperative pain score trends analyzed.
Mean time to return to work or regular activity, in days, reported by the patient. | Within the first 90 days after the surgery
  The time to return to work or regular activity after surgery as reported by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Seow-En, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Medina-Gallardo A, Curbelo-Pena Y, De Castro X, Roura-Poch P, Roca-Closa J, De Caralt-Mestres E. Is the severe pain after Milligan-Morgan hemorrhoidectomy still currently remaining a major postoperative problem despite being one of the oldest surgical techniques described? A case series of 117 consecutive patients. Int J Surg Case Rep. 2017;30:73-75. doi: 10.1016/j.ijscr.2016.11.018. Epub 2016 Nov 15. PMID 27960130
- [Background] Hetzer FH, Demartines N, Handschin AE, Clavien PA. Stapled vs excision hemorrhoidectomy: long-term results of a prospective randomized trial. Arch Surg. 2002 Mar;137(3):337-40. doi: 10.1001/archsurg.137.3.337. PMID 11888463
- [Background] Watkins AA, Johnson TV, Shrewsberry AB, Nourparvar P, Madni T, Watkins CJ, Feingold PL, Kooby DA, Maithel SK, Staley CA, Master VA. Ice packs reduce postoperative midline incision pain and narcotic use: a randomized controlled trial. J Am Coll Surg. 2014 Sep;219(3):511-7. doi: 10.1016/j.jamcollsurg.2014.03.057. Epub 2014 May 23. PMID 25081937
- [Derived] Seow-En I, Chen LRH, Zhao Y, Ng YY, Tan EK. Cryotherapy reduces pain post-hemorrhoidectomy (CYPHER): a randomized, controlled, superiority trial of intra-anal ice after surgery for grade III hemorrhoids. Ann Coloproctol. 2025 Dec;41(6):537-544. doi: 10.3393/ac.2025.00549.0078. Epub 2025 Dec 24. PMID 41486911